CLINICAL TRIAL: NCT03681600
Title: Observatory of the Quality of Surgical Procedures for Digestive Cancers: Pilot Project.
Brief Title: Observatory of the Quality of Surgical Procedures for Digestive Cancers
Acronym: Obchir
Status: Terminated | Type: Observational
Why Stopped: COVID 19
Sponsor: Moroccan Society of Surgery (Other)
Collaborators: Institut de Recherche sur le Cancer (Other Government); L'Ecole nationale supérieure d'informatique et d'analyse des systèmes (ENSIAS)(Mohammed V university in Rabat) (Unknown); Faculté des sciences de Rabat (Mohammed V university in Rabat) (Unknown); Stratance Consulting (Unknown)
Responsible Party: Sponsor
Other Study IDs: MoroccanSS
Record Dates: First submitted 2018-03-28; First posted 2018-09-24 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Digestive System Neoplasms; Surgery; Surgery--Complications; Quality of Health Care; Medical Audit
Keywords: audit; cancer; guidelines; ouctomes; survival; digestive cancer surgery
MeSH Terms: conditions — Digestive System Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgery for digestive cancers is managed according to quality standards, validated by the scientific community. Despite the diffusion of these standards through the benchmarks of good practice, the results of the surgery remain disparate.

In many countries, this "inequality of opportunity" has justified the establishment of quality assurance systems to measure the results of surgery for one or more localizations of digestive cancer.

These surgical audit experiments have shown a positive, rapid and cost-effective impact on complication rates, recurrence rates and overall survival even in the absence of interventional measures. The data collected also helped to improve the management of subgroups of patients usually excluded from clinical trials.

In Morocco, the National Cancer Prevention and Control Plan provides for the establishment of a quality assurance system with the introduction of a system for monitoring and evaluating the care of patients. This pilot project is part of this framework, for the group of patients who are candidates for surgery for digestive cancers.

ELIGIBILITY:
Inclusion Criteria:

* patients operated for a digestive cancer, proven or suspected, in a curative or palliative intent In elective situation: inclusion from surgery programming In emergent situation: inclusion no later than 72 hours after surgery
* Cancer proven or suspected in the following digestive tract: colon, appendix, anus, rectum, esophagus, stomach, eso-gastric junction, bile ducts, ampulla of Vater , pancreas, duodenum, small intestine and liver.
* Patient willing and able to agree to participate in the study

Exclusion Criteria:

* Patient whose surgical intervention is indicated for:

  * a condition that is not a digestive tract cancer, including whether retrospectively surgical exploration and / or histological examination reveals digestive localization cancer
  * proven or suspected cancer of non-digestive location
  * a proven or suspected cancer of peritoneal localization
* Patient whose surgical intervention is indicated for a progressive disease or a local recurrence proven or suspected of a digestive localization cancer having already been the resected (with the exception of situations of iterative liver resection for liver metastasis hepatic and recovery of the tumor bed after the discovery of vesicular cancer on cholecystectomy specimen)
* Patients whose intervention is for diagnostic purposes without any curative or palliative intention
* Patients whose surgery is a liver transplant
* Patients whose surgical intervention is local destruction (radiofrequency, microwaves) exclusively by percutaneous approach (without laparotomy or laparoscopy)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated for digestive cancer from 1st January 2018 to December 2020 in 4 moroccan surgical departments
Sampling Method: Non-Probability Sample
Enrollment: 1043 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
90-day Mortality rate | 90 days from surgery
  Death within 90 days of surgical procedure
90-day Complication rate | 90 days from surgery
  Defined with by Clavien-Dindo grade I to IV within90 days of surgical procedure
3-year Overall survival | from the date of operation to date of death from any cause, whichever came first, assessed up to 3 year
  Overall survival is defined as time from initiation to death of any cause within 3years of surgical procedure
3-year disease free survival | from operation until recurrence of tumor or death from any cause, whichever came first, assessed up to 3 years
  Disease free survival is defined as time from initiation to death of any cause within 3years of surgical procedure

SECONDARY OUTCOMES:
Treatment decisions made within multidisciplinary team meeting / tumour board | Prior to surgery
  For every localization
Availability/performance of CT chest, abdomen and pelvis scan performed for pre-operative staging | Prior to surgery
  For every localization

CONTACTS AND LOCATIONS:
Overall Officials: Amine Benkabbou, Pr, Study Director — Moroccan Society of Surgery; Raouf Mohsine, Pr, Principal Investigator — National institut of oncology; Abdelmalek Hrora, Pr, Principal Investigator — Moroccan Society of Surgery
Locations (4):
- Morocco (4):
  - National Institut of Oncology, Surgical oncology department, Rabat, Please Enter the State Or Province
  - Regional center of oncology, surgical department, Oujda
  - Ibn Sina Hospital, Surgical department A, Rabat
  - Ibn Sina Hospital, Surgical department C, Rabat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the project — https://sites.google.com/um5s.net.ma/observatoire